CLINICAL TRIAL: NCT03589144
Title: LC-MS / MS Adrenal Steroids Assayed on Dried Blot Spot for the Congenital Adrenal Hyperplasia Neonatal Screening: a Pilot, Multicenter, Prospective Study
Brief Title: LC-MS / MS Adrenal Steroids Assayed on Dried Blot Spot for the Congenital Adrenal Hyperplasia Neonatal Screening (SPECTROSPOT)
Acronym: SPECTROSPOT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17050J
Record Dates: First submitted 2018-06-06; First posted 2018-07-17 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Adrenal Hyperplasia, Congenital
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research uses the Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS / MS) technique on dried blot spot samples for the neonatal screening of congenital adrenal hyperplasia.

The main objective of this study is to demonstrate that this technique allow dosage of adrenal steroids on dried blot spot samples as efficiently and with the same sensitivity than the current technic on a cohort of 132 newborns aged 2 to 5 days, with a gestational age greater than or equal to 30 weeks of amenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 48 and 120 hours of life.
* Term of gestation: 30 to 41 weeks of gestation + 6 days
* weight at inclusion ≥ 1000 g
* non-opposition of the holders of parental authority

Exclusion Criteria:

* Patient who already had neonatal screening prior to inclusion.
* Patients whose health status contraindicates additional blood collection at the time of neonatal screening.
* Inability to give legal representatives of newborns informed information
* Minor Parents

Ages: 48 Hours to 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: National neonatal screening covers all newborns aged between 48 and 120 hours, regardless of birth term. Premature babies born before 30 weeks of amenorrhoea are cared for in specialized neonatal or intensive care units and are intensively monitored to rule out any risk of not diagnosing HCS in a child with it. This is why our study will be conducted on a newborn population with a birth term greater than 30 weeks of amenorrhoea.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient between the values of steroids assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term in neonates aged from 48 to 120 hours of life | 15 months
  Intra-class correlation coefficient between the values of 21 Deoxycortisol (21DF), 17hydroxyprogesterone (17OHP), pregnenolone, 17hydroxypregnenolone and cortisol assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term in neonates aged from 48 to 120 hours of life

SECONDARY OUTCOMES:
Study the difference between the levels of steroids assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates according to the term of birth (weeks) | 15 months
  Study the difference between the levels 21DF, 17OHP, pregnenolone, 17hydroxypregnenolone and cortisol assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the term of birth (weeks)
Study the difference between the levels of steroids assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates of life according to the mode of delivery (low or Caesarean section before work) | 15 months
  Study the difference between the levels 21DF, 17OHP, pregnenolone, 17hydroxypregnenolone and cortisol assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the mode of delivery (low or Caesarean section before work)
Study the difference between the levels of steroids assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates according to the presence or not of a corticotherapy antenatal. | 15 months
  Study the difference between the levels 21DF, 17OHP, pregnenolone, 17hydroxypregnenolone and cortisol assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the presence or not of a corticotherapy antenatal.
Study the difference between the levels of steroids assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the presence or not of non-maternal-fetal infection | 15 months
  Study the difference between the levels 21DF, 17OHP, pregnenolone, 17hydroxypregnenolone and cortisol assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the presence or not of non-maternal-fetal infection (chorioamnionitis, neonatal infection at the time of screening)
Study the difference between the levels of steroids assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the presence or not of newborn stress. | 15 months
  Study the difference between the levels 21DF, 17OHP, pregnenolone, 17hydroxypregnenolone and cortisol assayed by LC-MS / MS on dried blood spot and serum of preterm infants and full-term neonates aged from 48 to 120 hours of life according to the presence or not of newborn stress (septic shock and/or hypovolemic shock).

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle de périnatalité Service de néonatologie, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided